CLINICAL TRIAL: NCT00538252
Title: Parental Involvement, Extra-Familial Contexts and Prevention of Drug Use Risk
Brief Title: Parental Involvement and Children's Extra-Familial Contexts
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Daniel Shaw, Professor and Chair, University of Pittsburgh
Other Study IDs: involvementincontext; R01DA023245 (NIH); DA023245
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Prevention of Drug Abuse Risk
Keywords: drug use, antisocial behavior, early intervention, prevention
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Parental involvement has been shown to be a robust predictor of child conduct problems (CP) and drug use risk in childhood and adolescence, but relatively little attention has been paid to the role of parental involvement in relation to child problem behavior during the transition to school-age, when children are spending more time in school, after-care settings, and in the neighborhood. Concomitantly, as children transition from preschool to school-age, there is evidence to suggest that the quality and organization of schools, after-school care, and neighborhoods play an increasingly important role in the emergence of children's CP and drug use risk. Specifically, we will address: 1) the extent to which the quality of school environments, after-school care, and neighborhoods are associated with the emergence of CP during the early school-age period; 2) how parental involvement in the toddler and preschool period may be associated with parental involvement and monitoring in extra-familial contexts in the early school-age years; 3) how parental involvement in schools, after-care, and the neighborhood, may moderate relationships between extra-familial factors and children's CP; and 4) whether a parenting intervention can increase parental involvement in school, after-care, and neighborhood contexts and decrease risk of children's subsequent CP. These issues will be tested with an existing sample of 731 ethnically-diverse children from urban, suburban, and rural sites. As all families in the study were recruited based on the presence of sociodemographic, family, and child risk factors, the cohort of children are at high risk for displaying a persistent trajectory of clinically-meaningful CP and drug use risk. Thus, the study has the potential to fill a much-needed void on associations between extra-familial contexts and risk for early-starting CP and later problem behavior during the early school-age years. Equally critical, the study can provide data on the potential moderating influence of involved parenting, its malleability for families facing multiple adversities, and whether family-based interventions can make a difference for children facing multiple adversities.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled sample of 731 children recruited on the basis of prior screening for socioeconomic, family, and child risk factors at age 2

Exclusion Criteria:

* All children and families needed to have a child 2-3 years of age with multiple socioeconomic, family, and child risk factors.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 731 toddlers and their families followed from age 2 to 9 recruited on the basis of low socioeconomic status, and the presence of family (e.g., parental depression, drug use) and child (disruptive behavior) risk.
Sampling Method: Non-Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2007-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Achenbach Teacher Report Form | collected annually when children are ages 7 to 9 years old
  Teachers reports on over 100 items covering children's externalizing and internalizing problem behavior

SECONDARY OUTCOMES:
Parental Monitoring Inventory | Collected annually when children are ages 7 to 9
  Both children and parents report on the amount and quality of monitoring parents provide regarding their children's after-school activities

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Shaw, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Tein JY, Wang FL, Oro V, Kim H, Shaw D, Wilson M, Lemery-Chalfant K. The role of early intervention for adolescent mental health and polydrug use: Cascading mediation through childhood growth in the general psychopathology (p) factor. Dev Psychol. 2023 Aug;59(8):1484-1495. doi: 10.1037/dev0001543. Epub 2023 May 18. PMID 37199932